CLINICAL TRIAL: NCT06376188
Title: Improving Breaking Bad News in Pediatrics by Simulated Communication: The Prospective Randomized Controlled SimCom Study
Brief Title: Improving Breaking Bad News in Pediatrics by Simulated Communication
Acronym: SimCom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Jennifer Bettina Brandt; MD MSc, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1582/2021 SimCom
Record Dates: First submitted 2024-04-03; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Communication; End of Life; Pediatric ALL
Keywords: communication; pediatrics; palliative care; simulation; resuscitation; breaking bad news
MeSH Terms: conditions — Communication; Death; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): no communication training prior to simulation scenario
- Communication-Trained (Other): communication training prior to simulation scenario
  Interventions: Other: communication training

INTERVENTIONS:
Other: communication training — The intervention group received a communication training session prior to the prebriefing and familiarization of the scenario, including advice on how to improve communication skills as well as how to create an optimal setting for difficult medical conversations. This communication training session has been created on the basis of an in-depth literature research.(Brock et al., 2019; Chumpitazi et al., 2016; Collins et al., 2018; Grant et al., 2016; Tobler et al., 2014; Vaidya et al., 1999; Yuan et al., 2019)
  Arms: Communication-Trained

SUMMARY:
Breaking bad news, especially a death notice, is an essential part of the medical profes-sional communication. Being inadequately trained in those skills this may result in un-pleasant psychosocial consequences for everyone involved.

This prospective, single-center, randomized controlled trial evaluated the delivery of a death notice to simulation parents out of the perspective of these parents (professional actors), the participants (students) and by video analysis. The simulation patient has prior unexpectedly died during a simulated resuscitation. The intervention group broke the bad news after receiving a short communication

DETAILED DESCRIPTION:
Conversations about death and dying present discomfort for both healthcare professionals, patients and their families. These conversations, emotionally laden, pose lasting challenges and impact decision-making. Despite extensive medical training, physicians often lack adequate communication skills for such conversations, leading to frustration and distress. Delivering bad news, particularly in pediatrics, requires managing not only medical intricacies but also emotional impact. Communication skills, crucial for such scenarios, are typically developed over time through observation and practice, yet are often inadequately emphasized in medical training. Our study aimed to assess the impact of communication training on medical students delivering death notifications to simulation parents in pediatric simulation scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Medical students, enrolled at the Medical University of Vienna.
* Successful completion the mandatory basic life support training "Block 16" in the third year of medical training and
* Successful completion of the mandatory communication seminar "Ärztliche Gesprächsführung B" also in the third year of medical training.
* Obtained written informed consent.

Exclusion Criteria:

* quality of the obtained video recordings were unsatisfactory and not usable for analysis
* unmet inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
score by simulation parents | up to 1 hour after the simulation
  evaluation of breaking bad news by simulation parents, via a newly created questionnaire, measured in points, minimum score of zero points, maximum score of 69 points, the higher the score the better the outcome

SECONDARY OUTCOMES:
score by participants | up to 1 hour after the simulation
  self-evaluation of breaking bad news by participants, via a newly created questionnaire, measured in points, minimum score of zero points, maximum score of 63 points, the higher the score the better the outcome
score of video analysis | through study completion, an average of 1 year
  evaluation of breaking bad news by video raters, via a newly created questionnaire, measured in points, minimum score of zero points, maximum score of 270 points, the higher the score the better the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bettina Brandt, MD MSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babu TA. Breaking bad news in the paediatric ICU: need for ethical practice. Indian J Med Ethics. 2013 Oct-Dec;10(4):278-9. doi: 10.20529/IJME.2013.085. No abstract available. PMID 24152358
- [Background] Bittner-Fagan H, Davis J, Savoy M. Improving Patient Safety: Improving Communication. FP Essent. 2017 Dec;463:27-33. PMID 29210557
- [Background] Brock KE, Tracewski M, Allen KE, Klick J, Petrillo T, Hebbar KB. Simulation-Based Palliative Care Communication for Pediatric Critical Care Fellows. Am J Hosp Palliat Care. 2019 Sep;36(9):820-830. doi: 10.1177/1049909119839983. Epub 2019 Apr 11. PMID 30974949
- [Background] de Moura Villela EF, Bastos LK, de Almeida WS, Pereira AO, de Paula Rocha MS, de Oliveira FM, Bollela VR. Effects on Medical Students of Longitudinal Small-Group Learning about Breaking Bad News. Perm J. 2020;24:19.157. doi: 10.7812/TPP/19.157. Epub 2020 Feb 14. PMID 32097117
- [Background] Chumpitazi CE, Rees CA, Chumpitazi BP, Hsu DC, Doughty CB, Lorin MI. Creation and Assessment of a Bad News Delivery Simulation Curriculum for Pediatric Emergency Medicine Fellows. Cureus. 2016 May 1;8(5):e595. doi: 10.7759/cureus.595. PMID 27335708